CLINICAL TRIAL: NCT04702425
Title: A Phase Ib, Multicenter Study of VOB560 in Combination With MIK665 in Patients With Relapsed/Refractory Non-Hodgkin Lymphoma, Relapsed/Refractory Acute Myeloid Leukemia, or Relapsed/Refractory Multiple Myeloma.
Brief Title: VOB560-MIK665 Combination First in Human Trial in Patients With Hematological Malignancies (Relapsed/Refractory Non-Hodgkin Lymphoma, Relapsed/Refractory Acute Myeloid Leukemia, or Relapsed/Refractory Multiple Myeloma)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVOB560A12101; 2020-004691-18 (EudraCT Number)
Record Dates: First submitted 2020-12-02; First posted 2021-01-08 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Non-Hodgkin Lymphoma (NHL); Acute Myeloid Leukemia (AML); Multiple Myeloma (MM)
Keywords: Phase Ib, BHLRM, VOB560, MIK665, NHL, AML, MM, Bcl2, Mcl1
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Myeloid, Acute; Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- VOB560-MIK665 - Part 1a (Experimental): Part 1a - Patients with relapsed/refractory non-Hodgkin lymphoma and relapsed/refractory multiple myeloma administered VOB560 and MIK665 as an intravenous (IV) infusion.
  Interventions: Drug: VOB560; Drug: MIK665
- VOB560-MIK665 - Part 1b (Experimental): Part 1b - Patients with relapsed/refractory acute myeloid leukemia administered VOB560 and MIK665 as an intravenous (IV) infusion.
  Interventions: Drug: VOB560; Drug: MIK665
- VOB560-MIK665 - Part 2a (Experimental): Part 2a - Patients with relapsed/refractory multiple myeloma with at least 10 patients with 1q gain cytogenetic abnormality and 10 patients with high risk R/R MM as defined in (Sonneveld et al 2016) administered VOB560 and MIK665 as an intravenous (IV) infusion.
  Interventions: Drug: VOB560; Drug: MIK665
- VOB560-MIK665 - Part 2b (Experimental): Part 2b - Patients with relapsed/refractory non-Hodgkin lymphoma with at least 10 patients with double-hit (DH) lymphoma, based on the overall bad prognosis and limited therapeutic options for patients with DH NHL administered VOB560 and MIK665 as an intravenous (IV) infusion.
  Interventions: Drug: VOB560; Drug: MIK665
- VOB560-MIK665 - Part 2c (Experimental): Part 2c - Patients with relapsed/refractory acute myeloid leukemia venetoclax refractory or insensitive with at least 6 patients M5 as proposed by French-American-British (FAB) group, based on the observation that venetoclax resistance in AML M5 can be caused by up-regulation of MCL1 administered VOB560 and MIK665 as an intravenous (IV) infusion.
  Interventions: Drug: VOB560; Drug: MIK665
- VOB560-MIK665 - Part 2d (Experimental): Part 2d - Patients with relapsed/refractory acute myeloid leukemia venetoclax naive patients administered VOB560 and MIK665 as an intravenous (IV) infusion.
  Interventions: Drug: VOB560; Drug: MIK665

INTERVENTIONS:
Drug: VOB560 — Powder for concentrate for solution for infusion
  Other Names: S65487
Drug: MIK665 — Concentrate for solution for infusion
  Other Names: S64315

SUMMARY:
The purpose of the study was to identify doses and schedules of VOB560 and MIK665 that can be safely given and to learn if the combination can have possible benefits for patients with Non-Hodgkin lymphoma (NHL), Multiple Myeloma (MM) or Acute Myeloid Leukemia (AML).

VOB560 and MIK665 are selective and potent blockers respectively of the B-cell lymphoma 2 (BCL2) protein and of the myeloid cell leukaemia 1 (MCL1) protein, proteins that may protect tumor cells from undergoing cell death. VOB560 and MIK665 are designed to block the functions of the BCL2 and MCL1 proteins, so that the tumor cells that rely on these proteins undergo cell death.

Preclinical data suggest that concomitant treatment with VOB560 in combination with MIK665 induces robust anti-tumor activity.

DETAILED DESCRIPTION:
This was an open-label, non-randomized multi-center phase Ib dose-escalation study with dose expansion arms in four different patient populations. Patients received VOB560 in combination with MIK665 in a once a week (QW) schedule over 21 days cycle. Less frequent dosing schedules could be explored based on emerging data. Patients were to be treated until disease progression or unacceptable toxicities occurred.

The study included a dose escalation part (Part 1) and a dose expansion part (Part 2).

The following escalation arms were planned:

* Arm A: relapsed/refractory (R/R) NHL and R/R MM
* Arm B: R/R AML There were 4 expansion arms planned. However, the expansion part of the study was not initiated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of one of the following hematologic malignancies:

  * relapsed and/or refractory patients with non-Hodgkin lymphoma with radiographically measurable disease with a clearly demarcated nodal lesion at least 1.5 cm in its largest dimension or a target extra nodal lesion at least 1.0 cm in its largest dimension
  * relapsed and/or refractory patients with MM treated with at least 2 prior regimens, including an IMiD, a proteasome inhibitor proteasome inhibitor, and anti-CD38 antibody (if available) and not eligible for treatment with other regimens known to provide clinical benefit, as determined by the investigator.
  * relapsed and/or refractory patients with Acute Myeloid Leukemia (AML), pathologically confirmed diagnosis as defined by the WHO Classification and with ≥ 5% blasts in bone marrow. Following ≥ 1 prior therapies who have relapsed or exhibited refractory disease (primary failure) and are deemed by the investigator not to be candidates for standard therapy, including re-induction with cytarabine or other established therapeutic regimens for patients with AML (patients who are suitable for standard re-induction chemotherapy or hematopoietic stem cell transplantation and willing to receive it are excluded).
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* Patient must be a candidate for serial bone marrow aspirate and/or biopsy according to the institution's guidelines and be willing to undergo a bone marrow aspirate and/or biopsy at screening, during and at the end of therapy on this study.

Exclusion Criteria:

1. History of severe hypersensitivity reactions to any ingredient of study treatment and/or their excipients.
2. Systemic antineoplastic therapy (including cytotoxic chemotherapy, alpha-interferon, kinase inhibitors or other targeted small molecules, and toxin immunoconjugates) or any experimental therapy within 14 days or 5 half-lives, whichever is shorter, before the first dose of study treatment.
3. High-risk patients for Tumor Lysis Syndrome according to Cairo et al 2010 criteria or local guidelines.
4. Impaired cardiac function or clinically significant cardiac disease, or history or current diagnosis of ECG abnormalities indicating significant risk of safety including any of the following:

   1. Concomitant clinically significant cardiac arrhythmias, e.g. sustained ventricular tachycardia, and clinically significant second- or third-degree AV block without a pacemaker
   2. Any history of clinical important abnormalities in rhythm, conduction or morphology of resting ECG e.g. complete left bundle branch block, third degree heart block
   3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, significant hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age
   4. Resting QTcF ≥450 msec (male) or ≥460 msec (female) at pre-treatment
   5. Use of agents known to prolong the QT interval unless it can be permanently discontinued for the duration of study.
   6. Abnormal echocardiogram (ECHO) or multi-gated acquisition scan (MUGA) at baseline (left ventricular ejection fraction [LVEF] <50%)
   7. Symptomatic congestive heart failure (New York Heart Association ≥ 3)
   8. Findings observed in the baseline cardiac MRI that might reflect an increased risk for cardiac adverse events.
5. Use of hematopoietic colony-stimulating growth factors (e.g. G-CSF, GM-CSF, M-CSF), thrombopoietin mimetics or erythroid stimulating agents ≤ 2 weeks prior to start of study treatment. If thrombopoietin mimetics or erythroid stimulating agents were initiated more than 2 weeks prior to the first dose of study treatment and the patient is on a stable dose, they can be maintained.
6. For AML patients: Peripheral blast counts > 25,000 blasts / mm3. Patients can receive hydroxyurea to control the peripheral blast counts as long as hydroxyurea can be stopped at least 24 hours prior to obtaining PD biomarkers at screening/baseline. Hydroxyurea can be restarted after sampling if clinically indicated to control blasts prior to the start of study treatment markers.
7. For patients with R/R NHL and R/R MM:

   * Absolute Neutrophil count < 1.0 x 109/L
   * Platelets count < 50 x 109/ L
   * Hemoglobin < 8 g/dl
8. Autologous stem cell transplant within 3 months before the first dose of study treatment.
9. Patients who have undergone a prior allogeneic stem cell transplant before the first dose of study treatment.
10. History of or current interstitial lung disease or pneumonitis grade ≥ 2.
11. Impaired hepatic and renal function defined as:

    * Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 1.5 x upper limit of normal (ULN)
    * Bilirubin >1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
    * Creatinine clearance <50 mL/min (calculated using Cockroft-Gault formula, or measured).
12. Lipase >1.5 x ULN or serum amylase >1.5 x ULN and no history of pancreatitis.
13. Increased cardiac troponin above the manufacturer's 99th percentile upper reference limit for local assay at screening

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of AEs and SAEs, including changes in lab values, vital signs, and ECGs | at month 18
  Month 18 is assumed to be study end
Incidence of Dose Limiting Toxicities (DLTs) during the first cycle of treatment with VOB560 and MIK665 in combination | at month 18
  Month 18 is assumed to be study end
Frequency of dose interruptions | at month 18
  Month 18 is assumed to be study end
Frequency of dose reductions | at month 18
  Month 18 is assumed to be study end
Dose intensities | at month 18
  Month 18 is assumed to be study end

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | at month 18
  Month 18 is assumed to be study end As per European LeukemiaNet (ELN) 2017 for relapse/refractory (R/R) AML As per International Myeloma Working Group (IMWG) 2016 for R/R MM As per Lugano Classification 2014 for R/R NHL
Complete Response (CR) rate (and rate of CR or sCR in R/R MM) | at month 18
  Month 18 is assumed to be study end As per European LeukemiaNet (ELN) 2017 for relapse/refractory (R/R) AML As per International Myeloma Working Group (IMWG) 2016 for R/R MM As per Lugano Classification 2014 for R/R NHL
Best Overall Response (BOR) | at month 18
  Month 18 is assumed to be study end As per European LeukemiaNet (ELN) 2017 for relapse/refractory (R/R) AML As per International Myeloma Working Group (IMWG) 2016 for R/R MM As per Lugano Classification 2014 for R/R NHL
Duration Of Response (DOR) | at month 18
  Month 18 is assumed to be study end Month 18 is assumed to be study end As per European LeukemiaNet (ELN) 2017 for relapse/refractory (R/R) AML As per International Myeloma Working Group (IMWG) 2016 for R/R MM As per Lugano Classification 2014 for R/R NHL
Progression Free Survival (PFS) | at month 18
  Month 18 is assumed to be study end As per European LeukemiaNet (ELN) 2017 for relapse/refractory (R/R) AML As per International Myeloma Working Group (IMWG) 2016 for R/R MM As per Lugano Classification 2014 for R/R NHL
Area Under Curve (AUC) of VOB560 | At the end of Cycle 6 (each cycle is 21 days)
  PK parameter
Maximum Plasma Concentration (Cmax) ok VOB560 | At the end of Cycle 6 (each cycle is 21 days)
  PK parameter
Terminal elimination half-life (T1/2) of VOB560 | At the end of Cycle 6 (each cycle is 21 days)
  PK parameter
Clearance (CL) of VOB560 | At the end of Cycle 6 (each cycle is 21 days)
  PK parameter
Apparent volume of distribution (Vz) of VOB560 | At the end of Cycle 6 (each cycle is 21 days)
  PK parameter
Area Under Curve (AUC) of MIK665 | At the end of Cycle 6 (each cycle is 21 days)
  PK parameter
Maximum Plasma Concentration (Cmax) ok MIK665 | At the end of Cycle 6 (each cycle is 21 days)
  PK parameter
Terminal elimination half-life (T1/2) of MIK665 | At the end of Cycle 6 (each cycle is 21 days)
  PK parameter
Clearance (CL) of MIK665 | At the end of Cycle 6 (each cycle is 21 days)
  PK parameter
Apparent volume of distribution (Vz) of MIK665 | At the end of Cycle 6 (each cycle is 21 days)
  PK parameter

CONTACTS AND LOCATIONS:
Locations (9):
- Uni of TX MD Anderson Cancer Cntr UT MD Anderson Cancer Ctr, Houston, Texas, United States
- Novartis Investigative Site, Ghent, Belgium
- Novartis Investigative Site, HUS, Finland
- Novartis Investigative Site, Hong Kong, Hong Kong
- Novartis Investigative Site, Tel Aviv, Israel
- Novartis Investigative Site, Rozzano, MI, Italy
- Novartis Investigative Site, Sunto Gun, Shizuoka, Japan
- Novartis Investigative Site, Seoul, South Korea
- Novartis Investigative Site, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study results on Novartis clinical trials results database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18326
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2718